CLINICAL TRIAL: NCT05710991
Title: A Randomized Controlled Trial Examining the Impact of a Brief, Proactive, Cognitive Behavioural Therapy Versus Sleep Hygiene for Sleep Difficulties in Early Pregnancy
Brief Title: Brief Cognitive Behavioural Therapy for Insomnia Versus Sleep Hygiene for Sleep Difficulties in Early Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Sheryl Green, Associate Professor, Clinical Psychologist, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CBTI-SleepHygiene-RCT
Record Dates: First submitted 2023-01-13; First posted 2023-02-02 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Sleep Disturbance; Perinatal Anxiety; Perinatal Depression
MeSH Terms: conditions — Parasomnias | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Hygiene Workshop (Active Comparator): The Sleep Hygiene workshop contains psychoeducation on sleep hygiene and has been modified to target the transitions and concerns faced by perinatal individuals. Sleep hygiene is commonly utilized as a treatment for insomnia in general practice, with the information provided through verbal advice and a sleep hygiene info sheet. As such, the sleep hygiene protocol used in this study reflects standard care commonly offered to perinatal individuals outside of our specialized clinic.
  Interventions: Behavioral: Sleep Hygiene Workshop
- Cognitive Behavioural Therapy for Insomnia Workshop (Experimental): The Cognitive Behavioural Therapy (CBT) for Insomnia workshop contains empirically supported strategies for insomnia that have been modified to target the transitions and concerns faced by perinatal individuals. CBT is the first-line treatment for insomnia and promising research on CBT for insomnia specifically during pregnancy and postpartum is emerging.
  Interventions: Behavioral: Cognitive Behavioural Therapy for Insomnia Workshop

INTERVENTIONS:
Behavioral: Sleep Hygiene Workshop — Psychoeducation on the perinatal period and sleep difficulties including principles of sleep hygiene conducive environment for sleep, bedtime routine, food, beverage, and stimulant consumption, exercise
  Arms: Sleep Hygiene Workshop
Behavioral: Cognitive Behavioural Therapy for Insomnia Workshop — The CBT-I workshop group contains empirically supported strategies for insomnia modified to target the transitions and concerns faced by perinatal individuals. Content includes Sleep drive, stimulus control, sleep restriction, counter-arousal techniques, cognitive restructuring
  Arms: Cognitive Behavioural Therapy for Insomnia Workshop

SUMMARY:
Pregnant and postpartum individuals often have difficulty sleeping and these sleep problems can negatively impact both the parent and infant. Research suggests that pregnant individuals prefer non-medication-based treatment for their sleep difficulties but there is a lack of research on the success of sleep treatment during pregnancy. Currently, there are two main non-medical treatments for sleep difficulties available. The first, cognitive behavioural therapy (CBT), is the first treatment recommended for insomnia and has been found to successfully treat insomnia during pregnancy and the postpartum period. In addition, shortened sessions of CBT for insomnia have also been found to successfully reduce sleep difficulties. The second option is sleep hygiene education which is the most commonly offered treatment for sleep difficulties and has been found to improve sleep problems. The present study will compare the effectiveness of a CBT for insomnia group workshop to a Sleep Hygiene group workshop.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years
2. First, second, or third trimester of pregnancy (up to 34 weeks gestation) to allow for early/proactive benefit of sleep intervention.
3. Subjective difficulties with sleep (a score of 8 or higher on the Insomnia Severity Index)
4. Fluent in English.

Exclusion Criteria:

1. Severe depression/active suicidal ideation or psychotic
2. Unstable general medical condition
3. Current use of sleep aids or if taking a prescriptive medication, it remains stable in dose and type for study duration
4. a sleep disorder other than insomnia (e.g., restless leg syndrome).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Throughout the duration of the study (average of 10 months), change will be assessed at three timepoints: pre-treatment baseline (prior to 26 weeks gestation), post-treatment (up to 34 weeks gestation), and again at 12 weeks postpartum.
  The ISI is a 7-item self-report questionnaire that assesses the nature, severity, and impact of insomnia. Items are scored on a 5-point Likert scale ranging from 0 ('no problem') to 4 ('very severe problem') with higher scores reflecting greater insomnia severity. Total scores between 0-7 indicate an absence of insomnia; scores between 8-14 suggest sub-threshold insomnia; scores between 15-21 indicate moderate insomnia; and scores between 22-28 suggest severe insomnia. The ISI has demonstrated good psychometric properties.

SECONDARY OUTCOMES:
State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA). | Throughout the duration of the study (average of 10 months), change will be assessed at three timepoints: pre-treatment baseline (prior to 26 weeks gestation), post-treatment (up to 34 weeks gestation), and again at 12 weeks postpartum.
  The STICSA is a 21-item self-report scale that assesses cognitive and somatic components of anxiety. The STICSA is comprised of a state scale that measures individuals' current anxiety symptoms, and a trait scale that assesses one's proneness to anxiety, more generally. In the present study, only the trait scale of the STICSA will be used. Items are scored on a 4-point scale ranging from 1 ('not at all') to 4 ('very much so'). The STICSA has demonstrated excellent validity and reliability. A cut-off score of 43 or higher on the STICSA has been suggested for detecting a probable anxiety disorder. The STICSA has been validated for use in clinical samples of adults with anxiety disorders, although not explicitly in perinatal samples.
Edinburgh Postnatal Depression Scale (EPDS) | Throughout the duration of the study (average of 10 months), change will be assessed at three timepoints: pre-treatment baseline (prior to 26 weeks gestation), post-treatment (up to 34 weeks gestation), and again at 12 weeks postpartum.
  The EPDS is a 10-item self-report measure that assesses symptoms of depression during the perinatal period. Items are scored on a 4-point scale ranging from 0 to 3, with higher scores reflecting greater depressive symptomatology. The EPDS has demonstrated good sensitivity and specificity for a diagnosis of Major Depressive Disorder (MDD). Cut-off scores of 15 and 13 or higher have been suggested for detecting a probable diagnosis of MDD during pregnancy and the postpartum period, respectively.
Difficulties in Emotion Regulation Scale (DERS) | Throughout the duration of the study (average of 10 months), change will be assessed at three timepoints: pre-treatment baseline (prior to 26 weeks gestation), post-treatment (up to 34 weeks gestation), and again at 12 weeks postpartum.
  The DERS is a 36-item self-report scale designed to assess difficulties with emotion regulation. The DERS contains six subscales that measure: non-acceptance goals, impulse, awareness, strategies, and clarity. Items are rated on a 5-point Likert scale, ranging from 1 (almost never, 0-10%) to 5 (almost always, 91-100%), with higher scores reflecting greater difficulties regulating emotions. The DERS has demonstrated good internal consistency (α=0.86) and test-retest reliability (0.74).
Generalized Anxiety Disorder 7-Item Scale (GAD-7) | Throughout the duration of the study (average of 10 months), change will be assessed at three timepoints: pre-treatment baseline (prior to 26 weeks gestation), post-treatment (up to 34 weeks gestation), and again at 12 weeks postpartum.
  The GAD-7 is a 7-item self-report measure that assesses anxiety symptom severity over a previous two-week period. Items are measured on a 4-point scale ranging from 0 ('not at all') to 3 ('nearly every day'). A cut-off score of 10 or higher with sensitivity of 89% and specificity of 82% has been suggested for detecting a probable diagnosis of Generalized Anxiety Disorder. The GAD-7 has also been validated for use in perinatal samples.
Penn State Worry Questionnaire (PSWQ) | Throughout the duration of the study (average of 10 months), change will be assessed at three timepoints: pre-treatment baseline (prior to 26 weeks gestation), post-treatment (up to 34 weeks gestation), and again at 12 weeks postpartum.
  The PSWQ is a 16-item self-report measure that assesses the tendency to worry. Items are scored on a 5-point scale ranging from 1 ('not typical at all') to 5 ('very typical'), with higher scores reflecting greater pathological worry. A cut-off score of 62 or higher has been suggested for determining a probable GAD diagnosis. The PSWQ has demonstrated excellent internal consistency and validity across various populations and has been validated for use in perinatal samples.
Pre-Sleep Arousal Scale (PSAS) | Throughout the duration of the study (average of 10 months), change will be assessed at three timepoints: pre-treatment baseline (prior to 26 weeks gestation), post-treatment (up to 34 weeks gestation), and again at 12 weeks postpartum.
  The PSAS is a 16-item self-report measure that assesses one's state of arousal as they fall asleep. The measure consists of two subscales, one intended to measure cognitive arousal and the other somatic arousal. Participants are asked to describe how intensely they generally experience each cognitive and somatic symptom as they attempt to fall asleep in their own bedroom. Items are scored on a 5-point scale from 1 ('not at all') to 5 ('extremely), with subscale scores ranging from 8-40. Higher scores represent greater pre-sleep arousal.
PROMIS Anxiety Short-Form (PROMIS-A-SF) | Throughout the duration of the study (average of 10 months), change will be assessed at three timepoints: pre-treatment baseline (prior to 26 weeks gestation), post-treatment (up to 34 weeks gestation), and again at 12 weeks postpartum.
  The PROMIS Anxiety Short-Form is an 8-item self-report measure designed to assess anxious apprehension and hyperarousal. Participants rated the frequency of their symptoms on a 5-point scale ranging from 1 ('not at all') to 5 ('very much'), with higher scores representing greater anxiety. The measure was adapted to assess the frequency of symptoms in the past day rather than the past 7 days as used previously. The PROMIS Anxiety Short-Form has demonstrated good internal consistency (Cronbach's α = .93) and good psychometric properties.
PROMIS Depression Short-Form (PROMIS-D-SF) | Throughout the duration of the study (average of 10 months), change will be assessed at three timepoints: pre-treatment baseline (prior to 26 weeks gestation), post-treatment (up to 34 weeks gestation), and again at 12 weeks postpartum.
  The PROMIS Depression Short-Form is an 8-item self-report measure that assesses negative mood and negative views of self. Participants rated the frequency of their symptoms on a 5-point scale ranging from 1 ('not at all') to 5 ('very much'), with higher scores representing greater depression. The measure was adapted to assess the frequency of symptoms in the past day rather than the past 7 days as used previously. The PROMIS Depression Short-Form has demonstrated good internal consistency (Cronbach's α = .95) and good psychometric properties.
Consensus Sleep Diary (CSD). | Throughout the duration of the study (average of 10 months), change will be assessed at three timepoints: pre-treatment baseline (prior to 26 weeks gestation), post-treatment (up to 34 weeks gestation), and again at 12 weeks postpartum.
  The CSD was developed by a committee of experts with the aim of proposing a new improved and standardized sleep diary. This sleep diary will be filled out in the morning and includes questions such as (a) what time the participant went to bed, (b) what time they intended to sleep, (c) how long they were awake during the night, (d) what time they woke for the final time, (e) what time they got out of bed, and (f) how much sleep the participant got that night. From this data, we will derive time in bed, sleep onset latency, wakefulness after sleep onset, total sleep time, and sleep efficiency.
Polysomnography (PSG). | Throughout the duration of the study (average of 10 months), change will be assessed at three timepoints: pre-treatment baseline (prior to 26 weeks gestation), post-treatment (up to 34 weeks gestation), and again at 12 weeks postpartum.
  PSG recordings will be obtained using a device recording system that is self-applied at home. Portable PSG devices are primarily used for the screening of obstructive sleep apnea and growing research supports their use to evaluate sleep architecture and sleep quality. Standard recommendations suggest using PSG as a quantitative dependent measure in sleep research. Following these recommendations, PSG will be used for 2 nights to identify and quantify sleep-related breathing disturbances, periodic limb movements during sleep, and derive sleep measures (e.g., sleep onset latency, wakefulness after sleep onset, number of awakenings, total sleep time, terminal wakefulness, sleep efficiency).
Actigraphy watches. | Throughout the duration of the study (average of 10 months), change will be assessed at three timepoints: pre-treatment baseline (prior to 26 weeks gestation), post-treatment (up to 34 weeks gestation), and again at 12 weeks postpartum.
  Actigraphy watches are wrist-worn and battery-operated activity monitors that look similar to a small wristwatch. These devices are used to measure sleep and activity patterns and are typically used as an adjunctive measure in the diagnosis and treatment of insomnia to improve the reliability of self-report estimates of sleep. In this study, data collected from the actigraphy watches will be used to calculate objective measures of sleep such as sleep efficiency, total sleep time, time in bed, sleep onset latency, number of awakenings during the night, time awake after sleep onset, and terminal wakefulness.

OTHER OUTCOMES:
Sociodemographic Factors | Throughout the duration of the study (average of 10 months), change will be assessed at three timepoints: pre-treatment baseline (prior to 26 weeks gestation), post-treatment (up to 34 weeks gestation), and again at 12 weeks postpartum.
  Sociodemographic information collected will include participant's gender, age, ethnicity, marital status, education level, income level, parity, medical and delivery history, family psychiatric history, medication usage, and treatment history.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, West 5th Campus, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No